CLINICAL TRIAL: NCT07255001
Title: Monitoring Physical Function Changes in Patients With Pancreatic Ductal Adenocarcinoma: Potential for Better Understanding of Treatment Trajectory and Survival
Brief Title: Using Strength Tests to Better Understand How Pancreatic Cancer Affects Muscle Mass and Quality of Life
Acronym: PanFit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H25-00754
Record Dates: First submitted 2025-09-02; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC); Hand Grip Strength
Keywords: Pancreatic ductal adenocarcinoma (PDAC); Hand grip strength (HGS); Quality of Life (QOL); Body composition; Cachexia; Sarcopenia; Physical function; Skeletal muscle; Adipose tissue
MeSH Terms: conditions — Cachexia; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main Study Arm (Experimental): The study arm all participants are enrolled into. Participants will complete hand grip strength assessments and questionnaires.
  Interventions: Device: Hand grip strength assessments using a dynamometer

INTERVENTIONS:
Device: Hand grip strength assessments using a dynamometer — Squeeze a dynamometer with one hand to measure hand grip strength.

SUMMARY:
The goal of this clinical trial is to measure hand grip strength in adults with pancreatic ductal adenocarcinoma (PDAC). The main questions it aims to answer are:

* Is it feasible to measure hand grip strength as part of a clinic visit?
* Are changes in hand grip strength related to changes in body composition?
* Is hand grip strength related to a person's well-being?
* Is hand grip strength related to how a tumour responds to treatment?

Participants will squeeze a device with their hand to measure their hand grip strength and complete questionnaires about their well-being when they are seen in clinic for their regular medical care for PDAC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Histological and/or radiological diagnosis of resectable, non-resectable, or metastatic PDAC. For resectable PDAC, adjuvant setting only.
* ECOG performance status 0-2.
* Life expectancy greater than 6 months as judged by the investigator.
* Planned for treatment, either as part of routine care or in combination with an investigational agent within another study.
* Ability to hold a dynamometer with one hand.

Exclusion Criteria:

* Individuals with CT imaging performed outside of Vancouver, BC, Canada.
* Individuals who are unfit to undergo CT imaging of the third lumbar vertebra (L3).
* Individuals who are currently participating in a structured moderate intensity resistance training program.
* Individuals who are otherwise judged by the investigator to be unfit to proceed with this protocol.
* Unable to comply with study assessments and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of Participants with Hand Grip Strength (HGS) Measurements at 6 Months From Treatment Start Date | From the date anti-cancer therapy is initiated until the 6-month follow-up assessment.
  The percentage of participants with hand grip strength (HGS) test results at 6 months from treatment start date. Hand grip strength is measured in kilograms with a hand-held dynamometer.

SECONDARY OUTCOMES:
Frequency of Participants with Hand Grip Strength (HGS) Measurements at Study Baseline | At the time of the baseline assessment for the study.
  The percentage of participants with hand grip strength (HGS) test results at study baseline. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Frequency of Participants with Hand Grip Strength (HGS) Measurements at 3 Months From Treatment Start Date | From the date anti-cancer therapy is initiated until the 3-month follow-up assessment.
  The percentage of participants with hand grip strength (HGS) test results at 3 months from treatment start date. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Frequency of Participants with Hand Grip Strength (HGS) Measurements at 9 Months From Treatment Start Date | From the date anti-cancer therapy is initiated until the 9-month follow-up assessment.
  The percentage of participants with hand grip strength (HGS) test results at 9 months from treatment start date. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Frequency of Participants with Hand Grip Strength (HGS) Measurements at 12 Months From Treatment Start Date | From the date anti-cancer therapy is initiated until the 12-month follow-up assessment.
  The percentage of participants with hand grip strength (HGS) test results at 12 months from treatment start date. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Proportion of Participants with Sarcopenia Using CT Image Alone (Sarcopenia CT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The percentage of participants at each timepoint that meet the criteria for sarcopenia using the established definitions determined by CT image alone, namely the sex- and BMI-specific cut-off points developed by Caan et al. (2017).
Proportion of Participants with Sarcopenia Using Physical Function Alone (Sarcopenia P) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The percentage of participants at each timepoint that meet the criteria for sarcopenia using the definition of the Sarcopenia Definitions and Outcomes Consortium (SDOC) (Bhasin et al. 2020).
Proportion of Participants with Sarcopenia Using a Combination of CT Image and Physical Function (Sarcopenia COMB) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The percentage of participants at each timepoint that meet the criteria for sarcopenia using the definition by the European Working Group on Sarcopenia in Older Adults (EWGSOP2) (Cruz-Jentoft et al. 2019), which is supported by the Asian Working Group for Sarcopenia (Chen et al. 2019), and the Australian and New Zealand Society for Sarcopenia and Frailty Research (Zanker et al. 2023a, Zanker et al. 2023b).
Strength and Direction of the Relationship Between Hand Grip Strength (HGS) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in hand grip strength (HGS) for each unit of increase in skeletal muscle index (SMI). Hand grip strength is measured in kilograms with a hand-held dynamometer. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Hand Grip Strength (HGS) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in hand grip strength (HGS) for each unit of increase in skeletal muscle density (SMD). Hand grip strength is measured in kilograms with a hand-held dynamometer. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Hand Grip Strength (HGS) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in hand grip strength (HGS) for each unit of increase in skeletal muscle gauge (SMG). Hand grip strength is measured in kilograms with a hand-held dynamometer. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Hand Grip Strength (HGS) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in hand grip strength (HGS) for each unit of increase in visceral adipose tissue (VAT). Hand grip strength is measured in kilograms with a hand-held dynamometer. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Hand Grip Strength (HGS) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in hand grip strength (HGS) for each unit of increase in subcutaneous adipose tissue (SAT). Hand grip strength is measured in kilograms with a hand-held dynamometer. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Hand Grip Strength (HGS) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in hand grip strength (HGS) for each unit of increase in intermuscular adipose tissue (IMAT). Hand grip strength is measured in kilograms with a hand-held dynamometer. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Hand Grip Strength (HGS) and Progression-Free Survival (PFS) | From the date anti-cancer therapy is initiated until the date of clinical progression, withdrawal, date of death, or end of study, whichever comes first, assessed up to 26 months.
  The change in hand grip strength (HGS) for each unit of increase in progression-free survival (PFS). Hand grip strength is measured in kilograms with a hand-held dynamometer. Progression-free survival is the length of time from the first dose of treatment until the date of clinical progression.
Strength and Direction of the Relationship Between Hand Grip Strength (HGS) and Overall Survival (OS) | From the date anti-cancer therapy is initiated until the date of death or end of study, whichever comes first, assessed up to 26 months.
  The change in hand grip strength (HGS) for each unit of increase in overall survival (OS). Hand grip strength is measured in kilograms with a hand-held dynamometer. Overall survival is the length of time from the initiation of treatment that participants survive.
Strength and Direction of the Relationship Between Hand Grip Strength (HGS) and Objective Response Rate (ORR) | From the date of the baseline assessment scan until the date of clinical progression, withdrawal, date of death, or end of study, whichever comes first, assessed up to 26 months.
  The change in hand grip strength (HGS) for each unit of increase in objective response rate (ORR). Hand grip strength is measured in kilograms with a hand-held dynamometer. Objective response rate is the proportion of participants who have a complete or partial response to treatment.
Difference in Hand Grip Strength (HGS) Between Treatment Regimens | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The difference in the amount of hand grip strength (HGS) between participants receiving different treatment regimens. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Hand Grip Strength (HGS) and Tumour Stage | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in hand grip strength (HGS) for each unit of increase in tumour stage as defined by the American Joint Committee on Cancer (AJCC). Hand grip strength is measured in kilograms with a hand-held dynamometer. Tumour stage describes the extent of cancer growth and spread.
Strength and Direction of the Relationship Between Hand Grip Strength (HGS) and Tumour Grade | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in hand grip strength (HGS) for each unit of increase in tumour grade as defined by a four-tier grading system. Hand grip strength is measured in kilograms with a hand-held dynamometer. Tumour grade describes the appearance of cancer cells and their expected growth rate.
Difference in Hand Grip Strength (HGS) Between Sites of Metastasis | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The difference in the amount of hand grip strength (HGS) between participants with different sites of metastasis. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Global Health Status (QoL, per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the global health status from the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The global health status measure (QL2) ranges in score from 0 to 100 with higher scores indicating a higher quality of life. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Physical Functioning (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The physical functioning scale (PF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Role Functioning (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in role functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The role functioning scale (RF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Role functioning measures a person's ability to participate in daily life. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Emotional Functioning (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in emotional functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The emotional functioning scale (EF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Cognitive Functioning (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in cognitive functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The cognitive functioning scale (CF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Social Functioning (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in social functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The social functioning scale (SF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Fatigue (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in fatigue, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom scale for fatigue (FA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Nausea and Vomiting (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in nausea and vomiting, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom scale for nausea and vomiting (NV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Pain (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in pain, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom scale for pain (PA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Dyspnoea (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dyspnoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom item of dyspnoea (DY) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Insomnia (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in insomnia, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom item of insomnia (SL) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Appetite Loss (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in appetite loss, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom item of appetite loss (AP) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Constipation (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in constipation, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom item of constipation (CO) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Diarrhoea (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in diarrhoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom item of diarrhoea (DI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Financial Difficulties (per EORTC QLQ-C30) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in financial difficulties, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom item of financial difficulties (FI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Food Aversion (per EORTC QLQ-CAX24) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in food aversion, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom scale for food aversion (AV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Eating and Weight Loss Worry (per EORTC QLQ-CAX24) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating and weight loss worry, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom scale for eating and weight loss worry (EW) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Eating Difficulties (per EORTC QLQ-CAX24) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating difficulties, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom scale for eating difficulties (EAT) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Loss of Control (per EORTC QLQ-CAX24) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in loss of control, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom scale for loss of control (LC) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Physical Decline (per EORTC QLQ-CAX24) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical decline, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in hand grip strength (HGS). The symptom scale for physical decline (PHY) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Dry Mouth (per EORTC QLQ-CAX24) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dry mouth, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in hand grip strength (HGS). The single item measure of dry mouth (DM) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Indigestion/Heartburn (per EORTC QLQ-CAX24) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in indigestion/heartburn, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in hand grip strength (HGS). The single item measure of indigestion/heartburn (IND) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Forcing Self to Eat (per EORTC QLQ-CAX24) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in forcing self to eat, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in hand grip strength (HGS). The single item measure of forcing self to eat (FOR) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Inadequate Information (per EORTC QLQ-CAX24) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in a participant's perception of receiving inadequate information about their weight loss from their care team, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in hand grip strength (HGS). The single item measure of receiving inadequate information about weight loss (INF) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Index Value (per EuroQol EQ-5D-5L) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the Index Value from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in hand grip strength (HGS). In Canada, the Index Value ranges from -0.148 to 0.949 with larger and more positive numbers indicating better health. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Health Status (EQ-VAS per EuroQol EQ-5D-5L) and Hand Grip Strength (HGS) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the visual analogue scale (EQ-VAS) from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in hand grip strength (HGS). EQ-VAS ranges from 0 to 100 with larger scores indicating better health. Hand grip strength is measured in kilograms with a hand-held dynamometer.
Strength and Direction of the Relationship Between Global Health Status (QoL, per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the global health status from the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The global health status measure (QL2) ranges in score from 0 to 100 with higher scores indicating a higher quality of life. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Physical Functioning (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The physical functioning scale (PF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Role Functioning (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in role functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The role functioning scale (RF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Role functioning measures a person's ability to participate in daily life. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Emotional Functioning (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in emotional functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The emotional functioning scale (EF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Cognitive Functioning (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in cognitive functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The cognitive functioning scale (CF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Social Functioning (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in social functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The social functioning scale (SF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Fatigue (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in fatigue, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom scale for fatigue (FA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Nausea and Vomiting (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in nausea and vomiting, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom scale for nausea and vomiting (NV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Pain (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in pain, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom scale for pain (PA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Dyspnoea (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dyspnoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom item of dyspnoea (DY) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Insomnia (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in insomnia, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom item of insomnia (SL) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Appetite Loss (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in appetite loss, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom item of appetite loss (AP) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Constipation (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in constipation, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom item of constipation (CO) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Diarrhoea (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in diarrhoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom item of diarrhoea (DI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Financial Difficulties (per EORTC QLQ-C30) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in financial difficulties, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom item of financial difficulties (FI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Food Aversion (per EORTC QLQ-CAX24) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in food aversion, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom scale for food aversion (AV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Eating and Weight Loss Worry (per EORTC QLQ-CAX24) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating and weight loss worry, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom scale for eating and weight loss worry (EW) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Eating Difficulties (per EORTC QLQ-CAX24) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating difficulties, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom scale for eating difficulties (EAT) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Loss of Control (per EORTC QLQ-CAX24) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in loss of control, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom scale for loss of control (LC) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Physical Decline (per EORTC QLQ-CAX24) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical decline, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle index (SMI). The symptom scale for physical decline (PHY) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Dry Mouth (per EORTC QLQ-CAX24) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dry mouth, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle index (SMI). The single item measure of dry mouth (DM) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Indigestion/Heartburn (per EORTC QLQ-CAX24) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in indigestion/heartburn, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle index (SMI). The single item measure of indigestion/heartburn (IND) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Forcing Self to Eat (per EORTC QLQ-CAX24) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in forcing self to eat, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle index (SMI). The single item measure of forcing self to eat (FOR) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Inadequate Information (per EORTC QLQ-CAX24) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in a participant's perception of receiving inadequate information about their weight loss from their care team, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle index (SMI). The single item measure of receiving inadequate information about weight loss (INF) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Index Value (per EuroQol EQ-5D-5L) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the Index Value from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in skeletal muscle index (SMI). In Canada, the Index Value ranges from -0.148 to 0.949 with larger and more positive numbers indicating better health. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Health Status (EQ-VAS per EuroQol EQ-5D-5L) and Skeletal Muscle Index (SMI) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the visual analogue scale (EQ-VAS) from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in skeletal muscle index (SMI). EQ-VAS ranges from 0 to 100 with larger scores indicating better health. Skeletal muscle index estimates overall muscle mass by dividing skeletal muscle area (SMA) or skeletal muscle mass (SMM) by height squared. SMI is measured in cm^2/m^2 and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Global Health Status (QoL, per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the global health status from the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The global health status measure (QL2) ranges in score from 0 to 100 with higher scores indicating a higher quality of life. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Physical Functioning (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The physical functioning scale (PF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Role Functioning (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in role functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The role functioning scale (RF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Role functioning measures a person's ability to participate in daily life. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Emotional Functioning (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in emotional functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The emotional functioning scale (EF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Cognitive Functioning (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in cognitive functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The cognitive functioning scale (CF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Social Functioning (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in social functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The social functioning scale (SF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Fatigue (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in fatigue, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom scale for fatigue (FA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Nausea and Vomiting (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in nausea and vomiting, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom scale for nausea and vomiting (NV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Pain (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in pain, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom scale for pain (PA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Dyspnoea (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dyspnoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom item of dyspnoea (DY) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Insomnia (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in insomnia, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom item of insomnia (SL) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Appetite Loss (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in appetite loss, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom item of appetite loss (AP) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Constipation (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in constipation, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom item of constipation (CO) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Diarrhoea (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in diarrhoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom item of diarrhoea (DI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Financial Difficulties (per EORTC QLQ-C30) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in financial difficulties, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom item of financial difficulties (FI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Food Aversion (per EORTC QLQ-CAX24) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in food aversion, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom scale for food aversion (AV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Eating and Weight Loss Worry (per EORTC QLQ-CAX24) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating and weight loss worry, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom scale for eating and weight loss worry (EW) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Eating Difficulties (per EORTC QLQ-CAX24) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating difficulties, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom scale for eating difficulties (EAT) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Loss of Control (per EORTC QLQ-CAX24) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in loss of control, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom scale for loss of control (LC) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Physical Decline (per EORTC QLQ-CAX24) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical decline, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle density (SMD). The symptom scale for physical decline (PHY) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Dry Mouth (per EORTC QLQ-CAX24) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dry mouth, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle density (SMD). The single item measure of dry mouth (DM) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Indigestion/Heartburn (per EORTC QLQ-CAX24) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in indigestion/heartburn, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle density (SMD). The single item measure of indigestion/heartburn (IND) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Forcing Self to Eat (per EORTC QLQ-CAX24) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in forcing self to eat, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle density (SMD). The single item measure of forcing self to eat (FOR) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Inadequate Information (per EORTC QLQ-CAX24) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in a participant's perception of receiving inadequate information about their weight loss from their care team, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle density (SMD). The single item measure of receiving inadequate information about weight loss (INF) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Index Value (per EuroQol EQ-5D-5L) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the Index Value from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in skeletal muscle density (SMD). In Canada, the Index Value ranges from -0.148 to 0.949 with larger and more positive numbers indicating better health. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Health Status (EQ-VAS per EuroQol EQ-5D-5L) and Skeletal Muscle Density (SMD) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the visual analogue scale (EQ-VAS) from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in skeletal muscle density (SMD). EQ-VAS ranges from 0 to 100 with larger scores indicating better health. Skeletal muscle density measures muscle composition, which includes the amount of fat and non-fat tissue within the muscle. SMD is measured in Hausefield Units (HU) and is calculated from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Global Health Status (QoL, per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the global health status from the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The global health status measure (QL2) ranges in score from 0 to 100 with higher scores indicating a higher quality of life. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Physical Functioning (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The physical functioning scale (PF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Role Functioning (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in role functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The role functioning scale (RF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Role functioning measures a person's ability to participate in daily life. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Emotional Functioning (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in emotional functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The emotional functioning scale (EF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Cognitive Functioning (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in cognitive functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The cognitive functioning scale (CF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Social Functioning (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in social functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The social functioning scale (SF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Fatigue (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in fatigue, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom scale for fatigue (FA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Nausea and Vomiting (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in nausea and vomiting, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom scale for nausea and vomiting (NV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Pain (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in pain, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom scale for pain (PA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Dyspnoea (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dyspnoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom item of dyspnoea (DY) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Insomnia (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in insomnia, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom item of insomnia (SL) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Appetite Loss (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in appetite loss, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom item of appetite loss (AP) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Constipation (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in constipation, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom item of constipation (CO) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Diarrhoea (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in diarrhoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom item of diarrhoea (DI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Financial Difficulties (per EORTC QLQ-C30) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in financial difficulties, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom item of financial difficulties (FI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Food Aversion (per EORTC QLQ-CAX24) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in food aversion, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom scale for food aversion (AV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Eating and Weight Loss Worry (per EORTC QLQ-CAX24) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating and weight loss worry, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom scale for eating and weight loss worry (EW) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Eating Difficulties (per EORTC QLQ-CAX24) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating difficulties, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom scale for eating difficulties (EAT) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Loss of Control (per EORTC QLQ-CAX24) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in loss of control, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom scale for loss of control (LC) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Physical Decline (per EORTC QLQ-CAX24) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical decline, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The symptom scale for physical decline (PHY) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Dry Mouth (per EORTC QLQ-CAX24) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dry mouth, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The single item measure of dry mouth (DM) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Indigestion/Heartburn (per EORTC QLQ-CAX24) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in indigestion/heartburn, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The single item measure of indigestion/heartburn (IND) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Forcing Self to Eat (per EORTC QLQ-CAX24) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in forcing self to eat, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The single item measure of forcing self to eat (FOR) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Inadequate Information (per EORTC QLQ-CAX24) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in a participant's perception of receiving inadequate information about their weight loss from their care team, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in skeletal muscle gauge (SMG). The single item measure of receiving inadequate information about weight loss (INF) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Index Value (per EuroQol EQ-5D-5L) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the Index Value from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in skeletal muscle gauge (SMG). In Canada, the Index Value ranges from -0.148 to 0.949 with larger and more positive numbers indicating better health. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Health Status (EQ-VAS per EuroQol EQ-5D-5L) and Skeletal Muscle Gauge (SMG) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the visual analogue scale (EQ-VAS) from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in skeletal muscle gauge (SMG). EQ-VAS ranges from 0 to 100 with larger scores indicating better health. Skeletal muscle gauge is a measure of both skeletal muscle quantity and quality. SMG is calculated as the product of skeletal muscle index (SMI) and skeletal muscle density (SMD) and so is indirectly calculated from CT imaging of the third lumbar vertebra (L3). SMG is measured in Hausefield Units (HU)*cm^2/m^2.
Strength and Direction of the Relationship Between Global Health Status (QoL, per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the global health status from the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The global health status measure (QL2) ranges in score from 0 to 100 with higher scores indicating a higher quality of life. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Physical Functioning (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The physical functioning scale (PF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Role Functioning (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in role functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The role functioning scale (RF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Role functioning measures a person's ability to participate in daily life. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Emotional Functioning (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in emotional functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The emotional functioning scale (EF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Cognitive Functioning (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in cognitive functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The cognitive functioning scale (CF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Social Functioning (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in social functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The social functioning scale (SF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Fatigue (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in fatigue, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom scale for fatigue (FA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Nausea and Vomiting (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in nausea and vomiting, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom scale for nausea and vomiting (NV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Pain (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in pain, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom scale for pain (PA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Dyspnoea (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dyspnoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom item of dyspnoea (DY) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Insomnia (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in insomnia, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom item of insomnia (SL) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Appetite Loss (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in appetite loss, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom item of appetite loss (AP) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Constipation (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in constipation, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom item of constipation (CO) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Diarrhoea (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in diarrhoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom item of diarrhoea (DI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Financial Difficulties (per EORTC QLQ-C30) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in financial difficulties, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom item of financial difficulties (FI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Food Aversion (per EORTC QLQ-CAX24) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in food aversion, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom scale for food aversion (AV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Eating and Weight Loss Worry (per EORTC QLQ-CAX24) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating and weight loss worry, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom scale for eating and weight loss worry (EW) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Eating Difficulties (per EORTC QLQ-CAX24) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating difficulties, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom scale for eating difficulties (EAT) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Loss of Control (per EORTC QLQ-CAX24) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in loss of control, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom scale for loss of control (LC) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Physical Decline (per EORTC QLQ-CAX24) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical decline, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The symptom scale for physical decline (PHY) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Dry Mouth (per EORTC QLQ-CAX24) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dry mouth, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The single item measure of dry mouth (DM) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Indigestion/Heartburn (per EORTC QLQ-CAX24) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in indigestion/heartburn, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The single item measure of indigestion/heartburn (IND) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Forcing Self to Eat (per EORTC QLQ-CAX24) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in forcing self to eat, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The single item measure of forcing self to eat (FOR) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Inadequate Information (per EORTC QLQ-CAX24) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in a participant's perception of receiving inadequate information about their weight loss from their care team, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in visceral adipose tissue (VAT). The single item measure of receiving inadequate information about weight loss (INF) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Index Value (per EuroQol EQ-5D-5L) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the Index Value from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in visceral adipose tissue (VAT). In Canada, the Index Value ranges from -0.148 to 0.949 with larger and more positive numbers indicating better health. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Health Status (EQ-VAS per EuroQol EQ-5D-5L) and Visceral Adipose Tissue (VAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the visual analogue scale (EQ-VAS) from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in visceral adipose tissue (VAT). EQ-VAS ranges from 0 to 100 with larger scores indicating better health. Visceral adipose tissue is fat that is stored deep within the abdominal cavity and surrounds abdominal organs. VAT assesses the volume of fat in the body. VAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Global Health Status (QoL, per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the global health status from the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The global health status measure (QL2) ranges in score from 0 to 100 with higher scores indicating a higher quality of life. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Physical Functioning (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The physical functioning scale (PF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Role Functioning (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in role functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The role functioning scale (RF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Role functioning measures a person's ability to participate in daily life. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Emotional Functioning (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in emotional functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The emotional functioning scale (EF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Cognitive Functioning (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in cognitive functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The cognitive functioning scale (CF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Social Functioning (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in social functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The social functioning scale (SF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Fatigue (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in fatigue, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom scale for fatigue (FA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Nausea and Vomiting (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in nausea and vomiting, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom scale for nausea and vomiting (NV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Pain (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in pain, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom scale for pain (PA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Dyspnoea (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dyspnoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom item of dyspnoea (DY) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Insomnia (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in insomnia, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom item of insomnia (SL) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Appetite Loss (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in appetite loss, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom item of appetite loss (AP) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Constipation (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in constipation, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom item of constipation (CO) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Diarrhoea (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in diarrhoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom item of diarrhoea (DI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Financial Difficulties (per EORTC QLQ-C30) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in financial difficulties, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom item of financial difficulties (FI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Food Aversion (per EORTC QLQ-CAX24) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in food aversion, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom scale for food aversion (AV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Eating and Weight Loss Worry (per EORTC QLQ-CAX24) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating and weight loss worry, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom scale for eating and weight loss worry (EW) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Eating Difficulties (per EORTC QLQ-CAX24) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating difficulties, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom scale for eating difficulties (EAT) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Loss of Control (per EORTC QLQ-CAX24) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in loss of control, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom scale for loss of control (LC) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Physical Decline (per EORTC QLQ-CAX24) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical decline, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The symptom scale for physical decline (PHY) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Dry Mouth (per EORTC QLQ-CAX24) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dry mouth, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The single item measure of dry mouth (DM) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Indigestion/Heartburn (per EORTC QLQ-CAX24) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in indigestion/heartburn, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The single item measure of indigestion/heartburn (IND) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Forcing Self to Eat (per EORTC QLQ-CAX24) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in forcing self to eat, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The single item measure of forcing self to eat (FOR) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Inadequate Information (per EORTC QLQ-CAX24) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in a participant's perception of receiving inadequate information about their weight loss from their care team, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). The single item measure of receiving inadequate information about weight loss (INF) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Index Value (per EuroQol EQ-5D-5L) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the Index Value from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). In Canada, the Index Value ranges from -0.148 to 0.949 with larger and more positive numbers indicating better health. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Health Status (EQ-VAS per EuroQol EQ-5D-5L) and Subcutaneous Adipose Tissue (SAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the visual analogue scale (EQ-VAS) from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in subcutaneous adipose tissue (SAT). EQ-VAS ranges from 0 to 100 with larger scores indicating better health. Subcutaneous adipose tissue is the layer of fat located directly beneath the skin, between the dermis and muscles. SAT assesses fat distribution in the body. SAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Global Health Status (QoL, per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the global health status from the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The global health status measure (QL2) ranges in score from 0 to 100 with higher scores indicating a higher quality of life. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Physical Functioning (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The physical functioning scale (PF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Role Functioning (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in role functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The role functioning scale (RF2) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Role functioning measures a person's ability to participate in daily life. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Emotional Functioning (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in emotional functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The emotional functioning scale (EF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Cognitive Functioning (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in cognitive functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The cognitive functioning scale (CF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Social Functioning (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in social functioning, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The social functioning scale (SF) ranges from 0 to 100 with higher scores indicating a higher/healthy level of functioning. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Fatigue (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in fatigue, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom scale for fatigue (FA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Nausea and Vomiting (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in nausea and vomiting, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom scale for nausea and vomiting (NV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Pain (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in pain, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom scale for pain (PA) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Dyspnoea (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dyspnoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom item of dyspnoea (DY) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Insomnia (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in insomnia, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom item of insomnia (SL) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Appetite Loss (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in appetite loss, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom item of appetite loss (AP) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Constipation (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in constipation, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom item of constipation (CO) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Diarrhoea (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in diarrhoea, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom item of diarrhoea (DI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Financial Difficulties (per EORTC QLQ-C30) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in financial difficulties, as measured by the EORTC QLQ-C30 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom item of financial difficulties (FI) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Food Aversion (per EORTC QLQ-CAX24) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in food aversion, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom scale for food aversion (AV) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Eating and Weight Loss Worry (per EORTC QLQ-CAX24) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating and weight loss worry, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom scale for eating and weight loss worry (EW) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Eating Difficulties (per EORTC QLQ-CAX24) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in eating difficulties, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom scale for eating difficulties (EAT) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Loss of Control (per EORTC QLQ-CAX24) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in loss of control, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom scale for loss of control (LC) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Physical Decline (per EORTC QLQ-CAX24) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in physical decline, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The symptom scale for physical decline (PHY) ranges from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Dry Mouth (per EORTC QLQ-CAX24) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in dry mouth, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The single item measure of dry mouth (DM) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Indigestion/Heartburn (per EORTC QLQ-CAX24) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in indigestion/heartburn, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The single item measure of indigestion/heartburn (IND) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Forcing Self to Eat (per EORTC QLQ-CAX24) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in forcing self to eat, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The single item measure of forcing self to eat (FOR) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Inadequate Information (per EORTC QLQ-CAX24) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in a participant's perception of receiving inadequate information about their weight loss from their care team, as measured by the EORTC QLQ-CAX24 questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). The single item measure of receiving inadequate information about weight loss (INF) ranges in score from 0 to 100 with higher scores indicating a high level of symptomatology or problems. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Index Value (per EuroQol EQ-5D-5L) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the Index Value from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). In Canada, the Index Value ranges from -0.148 to 0.949 with larger and more positive numbers indicating better health. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).
Strength and Direction of the Relationship Between Health Status (EQ-VAS per EuroQol EQ-5D-5L) and Intermuscular Adipose Tissue (IMAT) | From the date anti-cancer therapy is initiated until the follow-up assessments at 3, 6, 9, and 12 months.
  The change in quality of life, as measured by the visual analogue scale (EQ-VAS) from the EuroQol EQ-5D-5L questionnaire, for each unit of increase in intermuscular adipose tissue (IMAT). EQ-VAS ranges from 0 to 100 with larger scores indicating better health. Intermuscular adipose tissue is fat that is located between muscle groups and underneath the deep fascia surrounding them. IMAT assesses the accumulation of fat in the body. IMAT is measured in cm^2 from CT imaging of the third lumbar vertebra (L3).

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared with other researchers.

REFERENCES:
- [Background] Armstrong V, Stretch C, Fitzgerald L, Gopaul A, McKinnon G, Koziak J, Kopciuk K, Brockton N, Bathe O. Characterizing cancer-associated myosteatosis: anatomic distribution and cancer-specific variability of low radiodensity muscle. JCSM Rapid Communications. 2021; 4(2):197-206. doi: 10.1002/rco2.46
- [Background] Song M, Zhang Q, Tang M, Zhang X, Ruan G, Zhang X, Zhang K, Ge Y, Yang M, Li Q, Li X, Liu X, Li W, Cong M, Wang K, Song C, Shi H. Associations of low hand grip strength with 1 year mortality of cancer cachexia: a multicentre observational study. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1489-1500. doi: 10.1002/jcsm.12778. Epub 2021 Sep 20. PMID 34545711
- [Background] Cheville A. Rehabilitation of patients with advanced cancer. Cancer. 2001 Aug 15;92(4 Suppl):1039-48. doi: 10.1002/1097-0142(20010815)92:4+3.0.co;2-l. PMID 11519031
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Wheelwright S, Darlington AS, Hopkinson JB, Fitzsimmons D, White A, Johnson CD. A systematic review of health-related quality of life instruments in patients with cancer cachexia. Support Care Cancer. 2013 Sep;21(9):2625-36. doi: 10.1007/s00520-013-1881-9. Epub 2013 Jun 25. PMID 23797577
- [Background] Cella D, Stone AA. Health-related quality of life measurement in oncology: advances and opportunities. Am Psychol. 2015 Feb-Mar;70(2):175-85. doi: 10.1037/a0037821. PMID 25730723
- [Background] Hagens ERC, Feenstra ML, van Egmond MA, van Laarhoven HWM, Hulshof MCCM, Boshier PR, Low DE, van Berge Henegouwen MI, Gisbertz SS. Influence of body composition and muscle strength on outcomes after multimodal oesophageal cancer treatment. J Cachexia Sarcopenia Muscle. 2020 Jun;11(3):756-767. doi: 10.1002/jcsm.12540. Epub 2020 Feb 25. PMID 32096923
- [Background] Caan BJ, Meyerhardt JA, Kroenke CH, Alexeeff S, Xiao J, Weltzien E, Feliciano EC, Castillo AL, Quesenberry CP, Kwan ML, Prado CM. Explaining the Obesity Paradox: The Association between Body Composition and Colorectal Cancer Survival (C-SCANS Study). Cancer Epidemiol Biomarkers Prev. 2017 Jul;26(7):1008-1015. doi: 10.1158/1055-9965.EPI-17-0200. Epub 2017 May 15. PMID 28506965
- [Background] Malietzis G, Aziz O, Bagnall NM, Johns N, Fearon KC, Jenkins JT. The role of body composition evaluation by computerized tomography in determining colorectal cancer treatment outcomes: a systematic review. Eur J Surg Oncol. 2015 Feb;41(2):186-96. doi: 10.1016/j.ejso.2014.10.056. Epub 2014 Nov 3. PMID 25468746
- [Background] Correa-de-Araujo R, Addison O, Miljkovic I, Goodpaster BH, Bergman BC, Clark RV, Elena JW, Esser KA, Ferrucci L, Harris-Love MO, Kritchevsky SB, Lorbergs A, Shepherd JA, Shulman GI, Rosen CJ. Myosteatosis in the Context of Skeletal Muscle Function Deficit: An Interdisciplinary Workshop at the National Institute on Aging. Front Physiol. 2020 Aug 7;11:963. doi: 10.3389/fphys.2020.00963. eCollection 2020. PMID 32903666
- [Background] Aleixo GFP, Shachar SS, Nyrop KA, Muss HB, Malpica L, Williams GR. Myosteatosis and prognosis in cancer: Systematic review and meta-analysis. Crit Rev Oncol Hematol. 2020 Jan;145:102839. doi: 10.1016/j.critrevonc.2019.102839. Epub 2019 Dec 20. PMID 31877534
- [Background] Mourtzakis M, Prado CM, Lieffers JR, Reiman T, McCargar LJ, Baracos VE. A practical and precise approach to quantification of body composition in cancer patients using computed tomography images acquired during routine care. Appl Physiol Nutr Metab. 2008 Oct;33(5):997-1006. doi: 10.1139/H08-075. PMID 18923576
- [Background] Alipour S, Kennecke HF, Woods R, Lim HJ, Speers C, Brown CJ, Gill S, Renouf DJ, Cheung WY. Body mass index and body surface area and their associations with outcomes in stage II and III colon cancer. J Gastrointest Cancer. 2013 Jun;44(2):203-10. doi: 10.1007/s12029-012-9472-4. PMID 23264206
- [Background] Zanker J, Sim M, Anderson K, Balogun S, Brennan-Olsen SL, Dent E, Duque G, Girgis CM, Grossmann M, Hayes A, Henwood T, Hirani V, Inderjeeth C, Iuliano S, Keogh J, Lewis JR, Lynch GS, Pasco JA, Phu S, Reijnierse EM, Russell N, Vlietstra L, Visvanathan R, Walker T, Waters DL, Yu S, Maier AB, Daly RM, Scott D. Consensus guidelines for sarcopenia prevention, diagnosis and management in Australia and New Zealand. J Cachexia Sarcopenia Muscle. 2023 Feb;14(1):142-156. doi: 10.1002/jcsm.13115. Epub 2022 Nov 9. PMID 36349684
- [Background] Cao A, Ferrucci LM, Caan BJ, Irwin ML. Effect of Exercise on Sarcopenia among Cancer Survivors: A Systematic Review. Cancers (Basel). 2022 Feb 3;14(3):786. doi: 10.3390/cancers14030786. PMID 35159052
- [Background] Zanker J, Sim M, Anderson K, Balogun S, Brennan-Olsen SL, Dent E, Duque G, Girgis CM, Grossmann M, Hayes A, Henwood T, Hirani V, Inderjeeth C, Iuliano S, Keogh J, Lewis JR, Lynch GS, Pasco JA, Phu S, Reijnierse EM, Russell N, Vlietstra L, Visvanathan R, Walker T, Waters DL, Yu S, Maier AB, Daly RM, Scott D. The Australian and New Zealand Society for Sarcopenia and Frailty Research (ANZSSFR) sarcopenia diagnosis and management task force: Findings from the consumer expert Delphi process. Australas J Ageing. 2023 Mar;42(1):251-257. doi: 10.1111/ajag.13164. Epub 2022 Dec 8. PMID 36480154
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Bhasin S, Travison TG, Manini TM, Patel S, Pencina KM, Fielding RA, Magaziner JM, Newman AB, Kiel DP, Cooper C, Guralnik JM, Cauley JA, Arai H, Clark BC, Landi F, Schaap LA, Pereira SL, Rooks D, Woo J, Woodhouse LJ, Binder E, Brown T, Shardell M, Xue QL, D'Agostino RB Sr, Orwig D, Gorsicki G, Correa-De-Araujo R, Cawthon PM. Sarcopenia Definition: The Position Statements of the Sarcopenia Definition and Outcomes Consortium. J Am Geriatr Soc. 2020 Jul;68(7):1410-1418. doi: 10.1111/jgs.16372. Epub 2020 Mar 9. PMID 32150289
- [Background] Groarke JD, Crawford J, Collins SM, Lubaczewski S, Roeland EJ, Naito T, Hendifar AE, Fallon M, Takayama K, Asmis T, Dunne RF, Karahanoglu I, Northcott CA, Harrington MA, Rossulek M, Qiu R, Saxena AR. Ponsegromab for the Treatment of Cancer Cachexia. N Engl J Med. 2024 Dec 19;391(24):2291-2303. doi: 10.1056/NEJMoa2409515. Epub 2024 Sep 14. PMID 39282907
- [Background] Dolly A, Dumas JF, Servais S. Cancer cachexia and skeletal muscle atrophy in clinical studies: what do we really know? J Cachexia Sarcopenia Muscle. 2020 Dec;11(6):1413-1428. doi: 10.1002/jcsm.12633. Epub 2020 Oct 14. PMID 33053604
- [Background] Tisdale MJ. Molecular pathways leading to cancer cachexia. Physiology (Bethesda). 2005 Oct;20:340-8. doi: 10.1152/physiol.00019.2005. PMID 16174873
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Vanhoutte G, van de Wiel M, Wouters K, Sels M, Bartolomeeussen L, De Keersmaecker S, Verschueren C, De Vroey V, De Wilde A, Smits E, Cheung KJ, De Clerck L, Aerts P, Baert D, Vandoninck C, Kindt S, Schelfhaut S, Vankerkhoven M, Troch A, Ceulemans L, Vandenbergh H, Leys S, Rondou T, Dewitte E, Maes K, Pauwels P, De Winter B, Van Gaal L, Ysebaert D, Peeters M. Cachexia in cancer: what is in the definition? BMJ Open Gastroenterol. 2016 Oct 18;3(1):e000097. doi: 10.1136/bmjgast-2016-000097. eCollection 2016. PMID 27843571
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Westbury LD, Beaudart C, Bruyere O, Cauley JA, Cawthon P, Cruz-Jentoft AJ, Curtis EM, Ensrud K, Fielding RA, Johansson H, Kanis JA, Karlsson MK, Lane NE, Lengele L, Lorentzon M, McCloskey E, Mellstrom D, Newman AB, Ohlsson C, Orwoll E, Reginster JY, Ribom E, Rosengren BE, Schousboe JT, Shiroma EJ, Harvey NC, Dennison EM, Cooper C; International Musculoskeletal Ageing Network. Recent sarcopenia definitions-prevalence, agreement and mortality associations among men: Findings from population-based cohorts. J Cachexia Sarcopenia Muscle. 2023 Feb;14(1):565-575. doi: 10.1002/jcsm.13160. Epub 2023 Jan 5. PMID 36604970
- [Background] Mueller TC, Burmeister MA, Bachmann J, Martignoni ME. Cachexia and pancreatic cancer: are there treatment options? World J Gastroenterol. 2014 Jul 28;20(28):9361-73. doi: 10.3748/wjg.v20.i28.9361. PMID 25071331
- [Background] Brown JC, Caan BJ, Prado CM, Cespedes Feliciano EM, Xiao J, Kroenke CH, Meyerhardt JA. The Association of Abdominal Adiposity With Mortality in Patients With Stage I-III Colorectal Cancer. J Natl Cancer Inst. 2020 Apr 1;112(4):377-383. doi: 10.1093/jnci/djz150. PMID 31355882
- [Background] Cespedes Feliciano EM, Lee VS, Prado CM, Meyerhardt JA, Alexeeff S, Kroenke CH, Xiao J, Castillo AL, Caan BJ. Muscle mass at the time of diagnosis of nonmetastatic colon cancer and early discontinuation of chemotherapy, delays, and dose reductions on adjuvant FOLFOX: The C-SCANS study. Cancer. 2017 Dec 15;123(24):4868-4877. doi: 10.1002/cncr.30950. Epub 2017 Sep 7. PMID 28881381
- [Background] Ali R, Baracos VE, Sawyer MB, Bianchi L, Roberts S, Assenat E, Mollevi C, Senesse P. Lean body mass as an independent determinant of dose-limiting toxicity and neuropathy in patients with colon cancer treated with FOLFOX regimens. Cancer Med. 2016 Apr;5(4):607-16. doi: 10.1002/cam4.621. Epub 2016 Jan 27. PMID 26814378
- [Background] Jung HW, Kim JW, Kim JY, Kim SW, Yang HK, Lee JW, Lee KW, Kim DW, Kang SB, Kim KI, Kim CH, Kim JH. Effect of muscle mass on toxicity and survival in patients with colon cancer undergoing adjuvant chemotherapy. Support Care Cancer. 2015 Mar;23(3):687-94. doi: 10.1007/s00520-014-2418-6. Epub 2014 Aug 28. PMID 25163434
- [Background] Yip C, Dinkel C, Mahajan A, Siddique M, Cook GJ, Goh V. Imaging body composition in cancer patients: visceral obesity, sarcopenia and sarcopenic obesity may impact on clinical outcome. Insights Imaging. 2015 Aug;6(4):489-97. doi: 10.1007/s13244-015-0414-0. Epub 2015 Jun 13. PMID 26070723
- [Background] Antoun S, Borget I, Lanoy E. Impact of sarcopenia on the prognosis and treatment toxicities in patients diagnosed with cancer. Curr Opin Support Palliat Care. 2013 Dec;7(4):383-9. doi: 10.1097/SPC.0000000000000011. PMID 24189893
- [Background] Prado CM, Baracos VE, McCargar LJ, Mourtzakis M, Mulder KE, Reiman T, Butts CA, Scarfe AG, Sawyer MB. Body composition as an independent determinant of 5-fluorouracil-based chemotherapy toxicity. Clin Cancer Res. 2007 Jun 1;13(11):3264-8. doi: 10.1158/1078-0432.CCR-06-3067. PMID 17545532
- [Background] Ngo-Huang AT, Parker NH, Xiao L, Schadler KL, Petzel MQB, Prakash LR, Kim MP, Tzeng CD, Lee JE, Ikoma N, Wolff RA, Javle MM, Koay EJ, Pant SD, Folloder JP, Wang X, Cotto AM, Ju YR, Garg N, Wang H, Bruera ED, Basen-Engquist KM, Katz MHG. Effects of a Pragmatic Home-based Exercise Program Concurrent With Neoadjuvant Therapy on Physical Function of Patients With Pancreatic Cancer: The PancFit Randomized Clinical Trial. Ann Surg. 2023 Jul 1;278(1):22-30. doi: 10.1097/SLA.0000000000005878. Epub 2023 Apr 7. PMID 37026453
- [Background] Lew D, Kamal F, Phan K, Randhawa K, Cornwell S, Bangolo AI, Weissman S, Pandol SJ. Epidemiologic risk factors for patients admitted with chronic pancreatitis and pancreatic ductal adenocarcinoma in the United States. World J Clin Oncol. 2022 Nov 24;13(11):907-917. doi: 10.5306/wjco.v13.i11.907. PMID 36483975